CLINICAL TRIAL: NCT07304297
Title: Impact of Intraoperative Tidal Volume on Surgical Parameters During Flexible Ureteroscopy
Brief Title: Effect of Tidal Volume on fURS Parameters
Acronym: TIDAL-fURS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarik Emre Sener (Other)
Responsible Party: Sponsor-Investigator, Tarik Emre Sener, Assistant Professor, Marmara University
Organization: Marmara University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAR.UAD.0026
Record Dates: First submitted 2025-11-30; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Urolithiasis; Tidal Volume; Flexible Ureteroscopy
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Tidal Volume (Active Comparator)
  Interventions: Procedure: Flexible Ureteroscopy
- Normal Tidal Volume (Placebo Comparator)
  Interventions: Procedure: Flexible Ureteroscopy

INTERVENTIONS:
Procedure: Flexible Ureteroscopy — Between October 2025 and December 2025, Patients who underwent fURS surgery in our clinic, with the surgical indication determined according to the EAU guidelines, were included in the study. Patients over 18 years of age with unilateral, single stones located in the upper or middle calyx or in the renal pelvis were included in the study. Patients with chronic obstructive pulmonary disease, pregnancy, a history of abdominal, retroperitoneal, or thoracic surgery, kidney anomalies, or stones located in the lower calyx were excluded.

SUMMARY:
The goal of this prospective clinical trial is to evaluate how intraoperative tidal volume settings affect surgical parameters and outcomes in adult patients undergoing flexible ureteroscopy (fURS) for kidney stones. The participant population includes patients over 18 years of age with unilateral, single renal stones located in the upper/middle calyx or renal pelvis.

This study aims to answer are:

Does intraoperative tidal volume influence operative time and surgical efficiency during fURS?

Does tidal volume affect laser energy use, lasing efficiency, stone-free rates, and complication rates (infection or bleeding)?

The investigators will compare two groups based on tidal volume recorded during anaesthesia:

Group 1: Low tidal volume (< 500 mL)

Group 2: Standard tidal volume (≥ 500 mL)

to determine whether tidal volume differences impact surgical performance and postoperative outcomes.

Participants will:

Undergo fURS performed under general anaesthesia with standard ASA monitoring, including ETCO₂ and TOF monitoring.

Have their respiratory parameters (tidal volume, peak airway pressure, PEEP, respiratory rate, ETCO₂) and surgical data (operative time, laser settings, fluoroscopy use, stone-free status) recorded during and after surgery.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years

Unilateral, single kidney stones located in the upper or middle calyx or in the renal pelvis

Exclusion Criteria:

Chronic obstructive pulmonary disease (COPD)

Pregnancy

History of abdominal, retroperitoneal, or thoracic surgery

Kidney anomalies

Stones located in the lower calyx

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-23 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Correlation Between Intraoperative Respiratory Parameters and Surgical Outcomes | 2 months
  Respiratory parameter measured:
  Tidal Volume (mL/kg)
  Measurement tool: Anaesthesia ventilator/monitoring system
  Unit: milliliters per kilogram (mL/kg)
  Surgical outcomes assessed:
  Stone-free rate (%), assessed by postoperative non-contrast CT scan
  Operative time (minutes), recorded from surgical logs
  Complications, graded using the Clavien-Dindo classification
  The objective is to determine the statistical correlation between tidal volume and each of these surgical outcomes.

SECONDARY OUTCOMES:
Correlation Between Intraoperative Respiratory Parameters and Seconder Outcomes | 2 months
  Operative time (minutes), recorded from surgical logs
  Surgical efficiency (stone volume / operative time, mm³/min)
  Laser time (seconds), recorded from laser console
  Laser energy used (Joules), recorded from laser console
  Lasing efficiency (stone volume / lasing time, mm³/sec)
  Complications, graded using the Clavien-Dindo classification
  Bleeding rate (%), incidence of significant intra- or postoperative bleeding
  Infection rate (%), incidence of postoperative urinary tract infection
  Length of hospital stay (days), total postoperative hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine Urology Department, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol